CLINICAL TRIAL: NCT03448835
Title: Neoadjuvant Capecitabine, Oxaliplatin, Docetaxel and Atezolizumab in Non-metastatic, Resectable Gastric and GE-junction Cancer: The PANDA Trial
Brief Title: Neoadjuvant Capecitabine, Oxaliplatin, Docetaxel and Atezolizumab in Resectable Gastric and GE-junction Cancer (PANDA)
Acronym: PANDA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N17PND
Record Dates: First submitted 2017-11-22; First posted 2018-02-28 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Stomach Cancer; Gastro Esophageal Junction Cancer
Keywords: short term immunotherapy; surgical resection; atezolizumab; capecitabine; oxaliplatin; docetaxel
MeSH Terms: conditions — Stomach Neoplasms | interventions — atezolizumab; Capecitabine; Oxaliplatin; Docetaxel

STUDY DESIGN:
Intervention Model Description: single group, open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- atezolizumab and chemotherapy (Experimental): 1 cycle of atezolizumab followed by 4 cycles atezolizumab, capecitabine, oxaliplatin and docetaxel
  Interventions: Drug: Atezolizumab; Drug: Capecitabine; Drug: Oxaliplatin; Drug: Docetaxel

INTERVENTIONS:
Drug: Atezolizumab — atezolizumab 1200 mg 5 cycles
  Other Names: MPDL3280A
Drug: Capecitabine — capecitabine 850 mg /m2 4 cycles
  Other Names: L01BC06
Drug: Oxaliplatin — oxaliplatin 100 mg/m2 4 cycles
  Other Names: L01XA03
Drug: Docetaxel — docetaxel 50 mg/m2 4 cycles
  Other Names: L01CD02

SUMMARY:
In this explorative study, patients with resectabel cancer of the stomach or stomach-oesophagealjunction cancer will receive neoadjuvant treatment.

The treatment will be 1 cyle atzolizumab monotherapy, followed by 4 cycle of atezolizumab and capecitabine, oxaliplatin and docetaxel.

DETAILED DESCRIPTION:
In this single-centre, open-label, monocenter study, the investigators will enroll 20 patients with resectable cancer of the stomach of GEJunction.

All patients will be treated with 1 cycle of atezolizumab monotherapy, followed by 4 cycles of combinationtherapy of atezolizumab, capecitabine, oxaliplatin and docetaxel, followed by surgery.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* patients age 18 and older
* primary resectable, histologically confirmed gastric or GEJ adenocarcinoma

Exclusion Criteria:

* no signs of distant metastases
* no active or history of autoimmune disease or immune deficiency
* no significant cardiovascular disease
* no major surgical procedure within 4 weeks prior to initiation of study treatment
* no current treatment with anti-viral therapy or HBV
* no pregnancy or breastfeeding
* no history of malignancy within 3 years prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03-07 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events following treatment (safety) | until 100 days after last patient last study drug treatment
  Adverse events will be assessed (according to CTC-AE v4.0) during treatment

SECONDARY OUTCOMES:
pathological tumor regression grade | Within 6 months after last patient inclusion
  determined using the Mandard tumor regression grading system

CONTACTS AND LOCATIONS:
Overall Officials: Myriam Chalabi, MD, Principal Investigator — Antoni van Leeuwenhoek
Locations (2):
- Netherlands (2):
  - Marieke van de Belt, Amsterdam
  - Catharina ziekenhuis, Eindhoven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verschoor YL, van de Haar J, van den Berg JG, van Sandick JW, Kodach LL, van Dieren JM, Balduzzi S, Grootscholten C, IJsselsteijn ME, Veenhof AAFA, Hartemink KJ, Vollebergh MA, Jurdi A, Sharma S, Spickard E, Owers EC, Bartels-Rutten A, den Hartog P, de Miranda NFCC, van Leerdam ME, Haanen JBAG, Schumacher TN, Voest EE, Chalabi M. Neoadjuvant atezolizumab plus chemotherapy in gastric and gastroesophageal junction adenocarcinoma: the phase 2 PANDA trial. Nat Med. 2024 Feb;30(2):519-530. doi: 10.1038/s41591-023-02758-x. Epub 2024 Jan 8. PMID 38191613
- [Derived] Chang X, Ge X, Zhang Y, Xue X. The current management and biomarkers of immunotherapy in advanced gastric cancer. Medicine (Baltimore). 2022 May 27;101(21):e29304. doi: 10.1097/MD.0000000000029304. PMID 35623069